CLINICAL TRIAL: NCT03888222
Title: A Randomized, Double Blind, Placebo-controlled Study to Evaluate the Impact of Bosutinib on Safety, Tolerability, Biomarkers and Clinical Outcomes in Dementia With Lewy Bodies (DLB)
Brief Title: Impact of Bosutinib on Safety, Tolerability, Biomarkers and Clinical Outcomes in Dementia With Lewy Bodies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Fernando Pagan MD, Associate Professor Of Neurology , Director of Movement Disorder Program, Medical Director of NPF COE at GUH , Fellowship Director, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#: STUDY00000017
Record Dates: First submitted 2019-03-13; First posted 2019-03-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease | interventions — bosutinib

STUDY DESIGN:
Intervention Model Description: We will evaluate the effects of 100 mg Bosutinib versus matching placebo taken daily by mouth for 12 weeks, followed by a 4 week wash-out period in individuals diagnosed with DLB. We will perform physiologically-based population pharmacokinetics (popPK) using a seamless random single dose (RSD) of Bosutinib, where participants (n=30) will be randomized to 3 groups (n=10) and take a single oral dose of 100mg, 200mg, Bosutinib or placebo (1;1;1) open label. Lumbar puncture will be performed between 1-4 hours after dosing. Participants will then be randomized double-blinded into 2 groups 1;1 using placebo(n=15) and 100mg (n=15) for 3 months.
  Randomization and Registration will be performed by an internet based randomization module. Randomization of the subjects to the 2 treatment groups will be performed in a stratified manner. The chance for randomization to the groups is 1:1 for placebo: 100 mg Bosutinib.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized by a Biostatistician by an internet based randomization module into two groups. The researchers include : Primary investigator , Sub-Investigators ,Clinical Coordinators, Nurse Practitioners , and Clinical Reseach unit staff.
  The investigators will be blinded to the dosage. Medications for any patient will be labeled by the CRU with a package medical identification number (Med. Id). A patient specific patient identification number (Pat. Id.) will be assigned to each patient. The investigator will have to note the Pat.Id on the designated medication package number after randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Thirty (30) participants will be recruited and randomized into 2 groups (arms) (1:1) .Fifteen (15) patients in group 1 will receive the matching placebo("sugar pill") one (1) capsule orally once daily for 3 months (90 days).
  Interventions: Drug: Placebo Oral Tablet
- 100 mg of Bosutinib (Active Comparator): Thirty (30) participants will be recruited and randomized into 2 groups (arms) (1:1) .Fifteen (15) patients in group 2 will receive the 100 mg of Bosutinib one (1) capsule orally once daily for 3 months (90 days).
  Interventions: Drug: Bosutinib Oral Tablet

INTERVENTIONS:
Drug: Placebo Oral Tablet — Fifteen (15) patients in group 1 will receive the matching placebo("sugar pill") one (1) tablet orally once daily for 3 months (90 days) .
  Other Names: Placebo
  Arms: Placebo
Drug: Bosutinib Oral Tablet — Fifteen (15) patients in group 1 will receive the 100 mg of Bosutinib one (1) tablet orally once daily for 3 months (90 days) .
  Other Names: Bosutinib(Bosulif®, SKI-606, Pfizer)
  Arms: 100 mg of Bosutinib

SUMMARY:
This study evaluates the effect of Bosutinib (Bosulif,Pfizer®) in the treatment of patients with Dementia with Lewy Bodies. Half participants will receive 100 mg of Bosutinib , while the other half will receive placebo.

DETAILED DESCRIPTION:
This proposal will evaluate the effects of Bosutinib (Bosulif, Pfizer®) treatment - an FDA-approved tyrosine kinase inhibitor that targets c-Abelson (Abl) and Src tyrosine kinases- in patients with DLB. Investigators have demonstrated safety and efficacy of this compound in pre-clinical animal models and others have shown similar benefits of Bosutinib on inflammation and neurotoxic protein clearance in neurodegeneration. Investigators have demonstrated that Bosutinib enters the brain (5% CSF:plasma ratio) and inhibits Abl at lower doses (5mg/kg) than the cancer dose (80mg/kg) in animals. Bosutinib also reduces the levels of neurotoxic proteins including alpha-synuclein, tau and beta-amyloid and improves motor and cognitive behavior in models of neurodegeneration. The use of Bosutinib is a novel strategy that promotes autophagy to clear neurotoxic protein aggregates in neurons. Bosutinib is FDA-approved for the treatment of chronic myelogenous leukemia (CML) at an oral dose of 400-600 mg daily. Based on our preclinical evidence, investigators used allometric conversion to extrapolate animal to human dose and estimated a human equivalent dose daily dose of 100mg Bosutinib in this clinical study to determine the safety and tolerability, pharmacokinetics and pharmacodynamics in patients with mild to moderate DLB.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Capable of providing informed consent and complying with study procedures. Subjects who are unable to provide consent may use a Legally Authorized Representative (LAR)
3. Age of 25-90 years, medically stable
4. Clinical diagnosis of DLB according to McKeith et al (7) with both dementia MoCA≥18 and Parkinsonian defined as bradykinesia in combination with rest tremor, rigidity or both UPDRS I-III ≤ 50 and UPDRS-III between 20-40.
5. Dementia and Parkinsonism must be present with at least one other symptom such as fluctuation, visual hallucinations or REM sleep behavioral disorder (RBD)
6. Abnormal DaTScan
7. Stable on Levodopa no more than 800mg daily, acetylcholinesterase inhibitors, dopamine agonists for at least 6 weeks
8. Stable on monoamine oxidase inhibitors (MOA-B) for at least 4 weeks before enrollment
9. Stable concomitant medical and/or psychiatric illnesses in the judgement of the PI
10. QTc interval 350-480 ms, inclusive
11. Participants must be willing to undergo LP at baseline and 3 months after treatment.

Exclusion Criteria:

1. Medical history of liver or pancreatic disease, GI ulcers and Chron's disease, kidney, GI, or blood problems
2. Abnormal liver function defined as AST and/or ALT > 100% the upper limit of the normal
3. Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal or proteinuria
4. History of HIV, clinically significant chronic hepatitis, or other active infection
5. hypokalemia, hypomagnesaemia, or long QT syndrome- QTc≥480 ms or concomitant drugs known to prolong the QTc interval and history of any cardiovascular disease, including myocardial infarction or cardiac failure, angina, arrhythmia
6. History or presence of significant cardiac conditions including: cardiovascular or cerebrovascular event (e.g. myocardial infarction, unstable angina, or stroke), congestive heart failure, first, second- or third-degree atrioventricular block, sick sinus syndrome, or other serious cardiac rhythm disturbances, any history of Torsade de Pointes.
7. Treatment with any of the following drugs at the time of screening or the preceding 30 days, and/or planned use over the course of the trial: Treatment with Class IA or III antiarrhythmic drugs (e.g. quinidine), treatment with QT prolonging drugs (www.crediblemeds.org)- excluding SSRIs (e.g. Citalopram, Escitalopram, Paroxetine, Sertraline, Duloxetine, Trazodone, etc.), Strong CYP3A4 inhibitors (including grapefruit juice). The concomitant use of strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole) must be avoided. Should treatment with any of these agents be required, therapy with Bosutinib should be interrupted. Anticoagulants, including Coumadin (warfarin), heparin, enoxaparin, daltiparin, xeralto, etc. St. John's Wort and the concomitant use of strong other CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital) must be avoided since these agents may reduce the concentration of Bosutinib
8. Females must not be lactating, pregnant or with possible pregnancy
9. Clinical signs indicating syndromes other than DLB including, Alzheimer's Disease (AD) idiopathic PD, corticobasal degeneration, supranuclear gaze palsy, multiple system atrophy, chronic traumatic encephalopathy, signs of frontal dementia, history of stroke, head injury or encephalitis, cerebellar signs, early severe autonomic involvement, Babinski sign
10. Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any active major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
11. Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving an investigational drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal or other systemic disease or laboratory abnormality.
12. Active neoplastic disease, history of cancer five years prior to screening, including breast cancer (history of skin melanoma or stable prostate cancer are not exclusionary)
13. Contraindications to LP: prior lumbosacral spine surgery, severe degenerative joint disease or deformity of the spine, platelets < 100,000, use of Coumadin/warfarin, or history of a bleeding disorder.
14. Must not be on any immunosuppressant medications
15. Must not be enrolled as an active participant in another clinical study.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability Go/NoGo (25% discontinuations) will be determined based on any emergent adverse events. | 3 Months
  We will determine safety and tolerability using the occurrence of adverse events (AEs) of interest, including myelosuppression, urinary, pancreatic and hepatic disorders, QTc prolongation as per Bosutinib IB.

SECONDARY OUTCOMES:
We will determine Bosutinib levels in CSF and plasma. | 3 Months
  We have demonstrated that Bosutinib enters the brain (5% CSF: plasma ratio) and inhibits Abl at lower doses (5mg/kg) than the cancer dose (80mg/kg) in animals. We predict that Bosutinib will be detected in the CSF. We will measure Bosutinib in both the CSF and Plasma and perform population pharmacokinetics.
We will determine changes in DLB related CSF and plasma biomarkers | 3 Months
  Plasma biomarkers include HVA, DOPAC, Abeta40/42, total tau, ptau231/181 and total and oligomeric alpha-synuclein. We expect Bosutinib to lower the levels of CSF markers of cell death, including neuron specific enolase (NSE), S100B and phosphorylated neurofilaments. We will also examine the effects of Bosutinib on other exploratory CSF and plasma inflammatory biomarkers, including triggering receptors on myeloid cells (TREM)-2, which is a potential risk factor for neurodegeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L Pagan, MD, Principal Investigator — Georgetown Univeristy
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hebron ML, Lonskaya I, Olopade P, Selby ST, Pagan F, Moussa CE. Tyrosine Kinase Inhibition Regulates Early Systemic Immune Changes and Modulates the Neuroimmune Response in alpha-Synucleinopathy. J Clin Cell Immunol. 2014 Sep 30;5:259. doi: 10.4172/2155-9899.1000259. PMID 25635231
- See also: https://sites.google.com/a/georgetown.edu/moussa-lab/lab-members — https://neurology.georgetown.edu/translational_neurotherapeutics